CLINICAL TRIAL: NCT06452823
Title: Cardiovascular Medicine Department of Second Affiliated Hospital of Jiaxing University
Brief Title: Efficacy and Safety of Catheter Ablation of Atrial Fibrillation in Patients With Thyroid Hormone Stabilization
Acronym: SQUIRREL
Status: Enrolling by invitation | Type: Observational
Sponsor: The Second Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Sponsor
Other Study IDs: CMDSAHJiaxing
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation and Flutter; Hyperthyroidism; Hypothyroidism
Keywords: Atrial Fibrillation and Flutter; Hyperthyroidism; Hypothyroidism; catheter radiofrequency ablation
MeSH Terms: conditions — Atrial Fibrillation; Hyperthyroidism; Hypothyroidism | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Combined Thyroid Dysfunction: Atrial catheter radiofrequency ablation for atrial fibrillation combined with patients requiring prior thyroid hormone abnormalities
  Interventions: Procedure: Catheter Ablation
- Uncomplicated thyroid dysfunction: Atrial catheter radiofrequency ablation for atrial fibrillation in patients with uncomplicated need for prior thyroid hormone abnormalities
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Procedure: Catheter Ablation — catheter radiofrequency ablation therapy for atrial fibrillation involves the use of ablative energy to destroy the cardiomyocytes at the opening of the pulmonary veins, which blocks the electrical conduction pathway between the pulmonary veins and the left atrium, so that atrial fibrillation no longer occurs.

SUMMARY:
Patients with hyperthyroidism or hypothyroidism are often combined with atrial fibrillation, but after the stabilization of thyroid hormone levels after treatment, the patients' atrial fibrillation still persists. Radiofrequency ablation of the atrial fibrillation as one of the treatment options for atrial fibrillation has been widely used in the clinic, and has significant efficacy in maintaining sinus rhythm, improving cardiac function, and improving the prognosis of patients. However, there is a lack of clinical monitoring data on radiofrequency ablation of atrial fibrillation in patients who have combined thyroid dysfunction and have stabilized their thyroid hormone levels after treatment.

DETAILED DESCRIPTION:
In patients recommended by guidelines for atrial catheter radiofrequency ablation of atrial fibrillation, catheter radiofrequency ablation was performed after exclusion of contraindications, and was observed and compared between patients with comorbid pre-existing thyroid hormone disorders and patients without comorbid atrial fibrillation after radiofrequency ablation:1: time to sexual rhythm maintenance: incidence of cardiac-related complications and incidence of noncardiac-related complications within 3 months and 1 year,2: walking distance on a six-minute walk test within 3 months,1 year, comparison of percent left ventricular ejection fraction, and comparison of left ventricular diastolic diameter at the time 3 months,1 year,.To comprehensively assess the efficacy and safety of catheterized radiofrequency ablation of atrial fibrillation in patients with comorbidities of prior thyroid hormone disorders.

ELIGIBILITY:
Inclusion Criteria:

Atrial Fibrillation Requiring Catheterized Radiofrequency Ablation （Class I Recommendation）

Exclusion Criteria:

Atrial Fibrillation Requiring Catheterized Radiofrequency Ablation Class I Recommendation With Coexisting Contraindications

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atrial Fibrillation Requiring Catheterized Radiofrequency Ablation Class I Recommendation Without Concurrent Contraindication
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation Recurrence of atrial fibrillation Recurrence of atrial fibrillation Recurrence of atrial fibrillation Recurrence of atrial fibrillation Recurrence of atrial fibrillation Recurrence of atrial fibrillation | 3 month and 1year after cardiac radiofrequency ablation
  Inability to maintain sinus rhythm, recurrent atrial fibrillation or atrial flutter
Postoperative heart-related complications | 3 month and 1year after cardiac radiofrequency ablation
  Cardiac perforation/cardiac tamponade Coronary artery stenosis/occlusion Pericarditis Atrial stiffness syndrome Coronary artery air embolism Pseudoaneurysm Severe pulmonary stenosis
Non-Cardiac Related Complications | 3 month and 1year after cardiac radiofrequency ablation
  Neurological Complications Asymptomatic cerebral embolism TIA Perioperative stroke Permanent phrenic nerve injury Digestive Complications Esophageal Injury Gastric Hyperdynamics Atrioesophageal Fistula Vascular Complications Hematoma Arteriovenous fistula Pseudoaneurysm Severe pulmonary stenosis

SECONDARY OUTCOMES:
6-minute walk test | 3 month and 1year after cardiac radiofrequency ablation
  Left atrial diastolic diameter
Left Atrial Internal Diameter | 3 month and 1year after cardiac radiofrequency ablation
  Left atrial anteroposterior and superior-inferior diameters
LVEF% | 3 month and 1year after cardiac radiofrequency ablation
  Per-beat output as a percentage of ventricular end-diastolic volume (cardiac preload)

OTHER OUTCOMES:
Thyroid hormone levels | 3 month and 1year after cardiac radiofrequency ablation
  hyperthyroidism Hypothyroidism A change in thyroid hormone status from stable to unstable.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Medicine Department of Second Affiliated Hospital of Jiaxing University, Jiaxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
no Plan to Share IPD